CLINICAL TRIAL: NCT05150314
Title: Comparative Study of the Hemorrhagic Risk in Patients Over 75 Years of Age Taking Enoxaparin at a Fixed Curative Dose of 4000 IU Twice a Day Versus at Dose / Weight Twice a Day as Part of the Treatment of Venous Thromboembolic Disease
Brief Title: Comparative Study of the Hemorrhagic Risk in Patients Over 75 Years of Age Taking Enoxaparin
Acronym: ENOX-VTD-H
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8426
Record Dates: First submitted 2021-11-25; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Venous Thromboembolic Disease
Keywords: Thrombophlebitis; Anticoagulant therapy; Enoxaparin; Venous Thromboembolic Disease
MeSH Terms: conditions — Thrombophlebitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Elderly subjects are at greater risk of thrombophlebitis than the general population, but also of bleeding when anticoagulant therapy is initiated.

Enoxaparin is one of the most widely used anticoagulants in the management of venous thromboembolism in the world.

Its use is not codified in the elderly, because too few studies have been carried out in people over 75 years old.

For several years, Enoxaparin in curative treatment has been administered at a reduced dosage of 4000 IU twice a day (and not at a standard dose of 100 IU / kg) at the Geriatrics center of the CRHU in Strasbourg with the clinical impression of a reduction the risk of serious bleeding without reduction in therapeutic efficacy in this very elderly population.

Confirmation of a reduction in the risk of bleeding at this dosage could be the start of a change in prescribing practices, towards a more suitable dosage in the elderly.

ELIGIBILITY:
Inclusion criteria:

* Subjects of age> = 75 years
* Having a weight> = 45kg for women and> = 57kg for men and a BMI <30, a GFR> 30 ml / min in Cockcroft-Gault, and having benefited from treatment with Enoxaparin for deep vein thrombosis and / or pulmonary embolism between 01/01/2000 to 11/30/2021.
* Subject having been informed by posting in the service and / or via the welcome booklet and not having expressed his opposition to the reuse of his data.

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* History of heparin-induced thrombocytopenia in the last 100 days,
* condition associated with a high risk of bleeding such as congenital or acquired blood pathology,
* a recent hemorrhagic stroke,
* a gastrointestinal ulcer,
* the presence of a malignant tumor at high risk of bleeding, recent surgery of the brain, spine or ophthalmology, known or suspected oesophageal varices, arteriovenous malformations, a vascular aneurysm or major intraspinal or intracerebral vascular anomalies.

Min Age: 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: - Subjects of age> = 75 years and having a weight> = 45kg for women and> = 57kg for men and a BMI <30, a GFR> 30 ml / min in Cockcroft-Gault, and having benefited from treatment with Enoxaparin for deep vein thrombosis and / or pulmonary embolism between 01/01/2000 to 11/30/2021.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-11-18 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04-18 (Estimated)

PRIMARY OUTCOMES:
Study of the risk of bleeding in patients over 75 years of age taking Enoxaparin at a fixed curative dose of 4000 IU twice a day | Files analysed retrospectively from January 01, 2000 to November 30, 2021 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Alexander BOUSSUGE, MD, Principal Investigator — Service de Gériatrie. Soins de Longue Durée - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Gériatrie. Soins de Longue Durée - Hôpitaux Universitaires de Strasbourg, Strasbourg, France